CLINICAL TRIAL: NCT03476330
Title: Quercetin Chemoprevention for Squamous Cell Carcinoma in Patients With Fanconi Anemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018-0073; 6353 (Other Grant/Funding Number: FDA Office of Orphan Products Development (OOPD))
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Fanconi Anemia; Squamous Cell Carcinoma
Keywords: Hematopoietic cell transplantation
MeSH Terms: conditions — Fanconi Anemia; Carcinoma, Squamous Cell | interventions — Quercetin; Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Quercetin (Experimental): All patients will be treated with oral quercetin.
  Interventions: Drug: Quercetin (dietary supplement)

INTERVENTIONS:
Drug: Quercetin (dietary supplement) — Quercetin will be administered twice daily at an adjusted dose based on weight for a maximum total daily dose of 4000mg/day. If the patient is 70 kg or more, the dose will automatically be assigned at the maximum dose of 4000mg/day.

SUMMARY:
Fanconi anemia (FA) is an autosomal recessive disease characterized by progressive bone marrow failure, variable congenital abnormalities and a predisposition to malignancy, particularly acute myeloid leukemia (AML) and squamous cell carcinoma (SCC). Improved transplant outcomes are modifying the natural history of Fanconi Anemia. Improved transplant survival, no radiation exposure, and almost no GVHD increases the importance of addressing later SCC even further. The investigators hypothesize that quercetin will prevent or delay the development of SCC and associated complications, there by ameliorating or delaying the need for potentially lethal treatment with chemotherapy and/or radiation therapy for the same.

Funding Source - FDA Office of Orphan Products Development (OOPD)

DETAILED DESCRIPTION:
Fanconi anemia (FA) is an autosomal recessive disease characterized by progressive bone marrow failure, variable congenital abnormalities and a predisposition to malignancy, particularly acute myeloid leukemia (AML) and squamous cell carcinoma (SCC). Currently, the only curative treatment option for the hematological complications of FA include hematopoietic cell transplantation (HCT). The investigators hypothesize that quercetin will prevent or delay the development of SCC and associated complications, there by ameliorating or delaying the need for potentially lethal treatment with chemotherapy and/or radiation therapy for the same.

This study is an open-label, single arm study. This study will enroll approximately 45 post-HCT patients with FA, and approximately 10 patients with FA without history of HCT. In both groups, patients with or without existing pre-malignant lesions or history of SCC will be allowed to participate, if they wish so and at the discretion of the PI. All patients will be treated with oral quercetin.

The investigators will determine the efficacy of Quercetin in reducing buccal micronuclei (a surrogate marker of DNA damage and susceptibility to squamous cell carcinoma due to genomic instability) in post-HCT patients with fanconi anemia (FA).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FA
* Able to take enteral medication
* Patients ≥2 years

Exclusion Criteria:

* Renal failure requiring dialysis
* Total bilirubin >3 mg/dl and/or SGPT >200 at time of enrollment
* Patients receiving digoxin therapy, who are unable to discontinue either treatment due to medical reasons
* Patients who are pregnant or breastfeeding or are at risk of pregnancy or fathering a baby and are unable to use acceptable methods of birth control during the length of the study
* Patients who have received quercetin supplementation or other antioxidants within the last 30 days
* Patients receiving radiation therapy, chemotherapy or immunotherapy for treatment of SCC.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Reduction of buccal micronuclei | Up to 30 months
  Efficacy of Quercetin in reducing buccal micronuclei

CONTACTS AND LOCATIONS:
Overall Officials: Parinda A Mehta, MD, Principal Investigator — Cincinnati Children's Hosptial Medical Center
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No